CLINICAL TRIAL: NCT02725645
Title: Influence of Different Backpack Loading Conditions on Neck and Lumbar Muscles Activity of Elementary School Children
Brief Title: Backpack Load and Spine Muscles Activity
Acronym: BLSMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Fernando Pessoa (Other)
Responsible Party: Principal Investigator, Sandra Rodrigues, Lecturer, University Fernando Pessoa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FCS-UFP-2016-03
Record Dates: First submitted 2016-03-21; First posted 2016-04-01 (Estimated); Results first posted 2019-10-28 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Child
Keywords: Surface electromyography; children; backpack

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy school children (Experimental): elementary school children will be presented with different backpack loading conditions
  Interventions: Other: loading conditions

INTERVENTIONS:
Other: loading conditions — Different backpack loading conditions 0%, 10%, 15% and 20% allocated randomly

SUMMARY:
The purpose of the present study is to analyze the influence of four backpack loading conditions (0, 10, 15 and 20% of body weight) on the electromyographic activity of the neck and lumbar muscles of elementary school children.

DETAILED DESCRIPTION:
Elementary school children participated in the present study, between the ages of 6 and 10. Bilateral sternocleidomastoid, rectus abdominis and erector spinae muscles activity were recorded using surface electromyography (sEMG), while tested for the effect of four randomized backpack loading conditions.

ELIGIBILITY:
Inclusion Criteria:

* children with tutor consent

Exclusion Criteria:

* children with cognitive impairment

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2014-06; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Rodrigues, MSc, Mphil, Principal Investigator — University Fernando Pessoa

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: elementary school children, male and female, with no history of spine problems. Tutors provided legal authorization.
Groups:
- Healthy School Children: Participants had to stand, using backpacks with different load conditions, while being monitored with emg.
Period: Overall Study
Arm/Group | Healthy School Children
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Healthy School Children: Participants had to stand with different backpack loading conditions.
Arm/Group | Healthy School Children
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.93 (0.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 5
Region of Enrollment [Number; unit: participants]
  Portugal | 14

OUTCOME MEASURES:

1. Primary Outcome: Muscle Activity as a Measure of Route Mean Square
Description: EMG signals were initially filtered with a Notch Filter of 50hz, due to the DC power line, using MATLAB 7.11 (v.2010). The signal was then detrended, converted into millivolts and normalized. the normalized signal was then used to calculate the route mean square.
Time Frame: one year
Measure: Mean (Standard Deviation); unit: milivolts
Groups:
- Healthy School Children: 14 elementary school children participated in the study, 9 female and 5 male.
Arm/Group | Healthy School Children
Number analyzed (Participants) | 14
milivolts
  left lumbar erector spinae at 0% of body weight | 13.96 (8.45)
  left lumbar erector spinae at 10% of body weight | 10.70 (7.31)
  left lumbar erector spinae at 15% of body weight | 10.85 (7.47)
  left lumbar erector spinae at 20% of body weight | 9.28 (5.47)
  Right lumbar erector spinae at 0% of body weight | 13.36 (8.73)
  Right lumbar erector spinae at 10% of body weight | 9.20 (7.47)
  Right lumbar erector spinae at 15% of body weight | 7.19 (3.67)
  Right lumbar erector spinae at 20% of body weight | 6.55 (2.91)
  Left cervical erector spinae at 0% of body weight | 8.56 (4.41)
  Left cervical erector spinae at 10% of body weight | 7.66 (2.43)
  Left cervical erector spinae at 15% of body weight | 8.69 (3.15)
  Left cervical erector spinae at 20% of body weight | 9.85 (4.50)
  Right cervical erector spinae at 0% of body weight | 7.77 (2.89)
  Right cervical erec spinae at 10% of body weight | 8.91 (3.81)
  Right cervical erec spinae at 15% of body weight | 9.32 (3.28)
  Right cervical erec spinae at 20% of body weight | 11.10 (3.67)
  Left Rectus Abdominis at 0% of body weight | 3.35 (0.29)
  Left Rectus Abdominis at 10% of body weight | 3.68 (0.60)
  Left Rectus Abdominis at 15% of body weight | 4.27 (1.77)
  Left Rectus Abdominis at 20% of body weight | 4.03 (1.16)
  Right Rectus Abdominis at 0% of body weight | 3.64 (0.32)
  Right Rectus Abdominis at 10% of body weight | 3.88 (0.29)
  Right Rectus Abdominis at 15% of body weight | 4.94 (2.58)
  Right Rectus Abdominis at 20% of body weight | 4.54 (1.50)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Participants were screened for any discomfort related to the use of surface emg electrodes and monitored for any possible dizziness.
Arm/Group | Healthy School Children
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes